CLINICAL TRIAL: NCT02630888
Title: Efficacy of the Combination of Memantine in the Treatment of Bipolar Disorder (Type I) Nonresponders or Partial Responders Young Patients to Previous Combination Therapy of Quetiapine Plus Lithium or Quetiapine Plus Aripiprazole
Brief Title: Efficacy of Memantine add-on in the Treatment of Bipolar Disorder (Type I) Nonresponders or Partial Responders Patients
Acronym: ARIQUELI-ME
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Ricardo Alberto Moreno, M.D., Ph.D., Affective disorders program (GRUDA), University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MORENO-2015
Record Dates: First submitted 2015-12-02; First posted 2015-12-15 (Estimated); Last update posted 2019-10-03 (Actual); Status verified 2019-10

CONDITIONS: Bipolar Disorder
Keywords: Bipolar Disorder; Memantine; Lithium; Aripiprazole; Quetiapine; Central Nervous System Agents; Therapeutic Uses; Pharmacologic Actions; Psychotropic Drugs; Cognitive effect of drugs
MeSH Terms: conditions — Bipolar Disorder | interventions — Memantine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Memantine (Active Comparator): Patients randomized to this group will receive a dose of 15 mg / day of memantine during the first week (V0); all have the dose of memantine increased on the second week (V1) at the dose of 30 mg / day (in two divided doses of 15 mg).
  Interventions: Drug: Memantine
- Placebo (Placebo Comparator): Patients randomized to this group will receive a unit dosage identical to that contains 15 mg of memantine during the first week (V0); all have the dose of the placebo (similar to memantine) increased on the second week (V1) in two divided doses of a unit dosage identical to that contains 15 mg of memantine.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Memantine — Memantine association in the treatment of young patients with Bipolar I Disorder, partial responders or non-responders to the combination of (quetiapine + lithium) or (quetiapine + aripiprazole) from the ARIQUELI study.
  Other Names: Namenda; Ebixa
  Arms: Memantine
Drug: Placebo — Patients randomized to this group will receive a unit dosage identical to that contains 15 mg of memantine during the first week (V0); all have the dose of the placebo (similar to memantine) increased on the second week (V1) in two divided doses of a unit dosage identical to that contains 15 mg of memantine
  Other Names: Non active drug
  Arms: Placebo

SUMMARY:
The main goal of this study is evaluate the efficacy of memantine association on the treatment with a previous combination of two drugs, including quetiapine with lithium or quetiapine with aripiprazole in young patients with bipolar disorder type 1 non-responders or partial responders to that combination of drugs and evaluate the impact of this association at the cognitive functioning of the patients.

DETAILED DESCRIPTION:
Current evidence suggests that deregulation of brain glutamatergic neurotransmission is involved in the pathophysiology of bipolar disorder and that drugs that intervene in this transmission may be therapeutic weapons in addressing the symptoms and cognitive deficits of this pathology. Among these drugs, particularly memantine is a strong candidate in view of their efficacy in antagonizing N-methyl-D-aspartate (NMDA) receptors, and their good safety and tolerability profile. The principal aim of this study is to evaluate the efficacy of memantine association with treatment with a combination of two drugs, including quetiapine with lithium and quetiapine with aripiprazole in young patients with bipolar disorder type 1 non-responders or partial responders and evaluate the impact of this association cognitive functioning of patients. An experimental study, randomized, double-blind, bipolar patients with type 1, of both sexes, aged 18 to 40, ambulatory or hospitalized, at any stage of the disease, seeking treatment in the Mood Disorders Program (GRUDA) of Institute os Psychiatry (IPq) of Sao Paulo University (FMUSP). Patients will come from ARIQUELI Project (Missio, G. et al, 2013 submitted Trial registration - ClinicalTrials.gov Identifier:. NCT01710163).

The study will be conducted in two stages: I - initial administration of memantine or placebo for 8 weeks; II - Maintenance administration for more 4 months.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1) Partial responders or non-responders (HAM-D score > 7 points and/or YMRS > 9 points) in the ARIQUELI Study (after quetiapine + lithium or quetiapine + aripiprazole combination).
* EXCLUSION CRITERIA:

  1. Patients with Schizophrenia, Schizoaffective Disorder or Mental Retardation (Intellectual Quotient Total less than 90);
  2. Patients with severe, unstable diseases, including kidney disease, gastroenterology, respiratory, cardiovascular, endocrine, neurological, immunological or haematological;
  3. Hypo or hyperthyroidism uncorrected;
  4. Angle-closure glaucoma;
  5. Changes in blood coagulation or use of regular anticoagulants;
  6. Patients with serious risk of suicide (according to clinical criteria and / or score> = 4 in the HAM-D item suicide) may participate in the study only in inpatients;

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 44 (Estimated)
Dates: Start 2014-08 (Actual); Primary Completion 2020-04 (Estimated); Study Completion 2020-09 (Estimated)

PRIMARY OUTCOMES:
Memantine efficacy in stabilizing mood | 8 weeks
  The primary outcome measure is to evaluate the memantine efficacy of the combination at 30 mg / day in stabilizing mood to therapy of young patients with Bipolar Disorder (type I) non-responders or partial responders to quetiapine combination with lithium or with aripiprazole from the ARIQUELI study. The definitions of the outcomes are:
  * Partial response: between 26% and 49% reduction from the baseline to the type of index episode (mania, mixed episode, depression), without further worsening of the opposite pole;
  * Response: ≥ 50% reduction from the baseline to the type of index episode (mania, mixed episode, depression) without further worsening of the opposite pole;
  * Remission: the used remission score is less than or equal to 9 of Young Mania Rating Scale (YMRS), equal or lower to 7 in Hamilton Depression Rating Scale (HAMD-21) reduction equal to or greater than 75% the inclusion scores in the study.

SECONDARY OUTCOMES:
Memantine impact in the cognitive functioning | 24 weeks (6 months)
  Improvement in the neuropsychological tests from baseline until the last observation carried forward in both groups (memantine x placebo).

CONTACTS AND LOCATIONS:
Overall Officials: Ricardo A. Moreno, MD, PhD, Study Director — Sao Paulo University
Locations (1):
- Institute of Psychiatry, University of Sao Paulo, São Paulo, Brazil